CLINICAL TRIAL: NCT00178516
Title: Vitamin E and Male Infertility
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Mae Stone Goode Foundation (Other)
Responsible Party: Vivian LEwis, MD, UNiversity of Rochester Medical Center
Other Study IDs: RSRB 10160
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Male Infertility
Keywords: male; infertility
MeSH Terms: conditions — Infertility, Male; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, semen
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: behavior, procedure

SUMMARY:
The goal of this study is to determine whether there is a correlation between the levels of Vitamin E in sperm and sperm DNA fragmentation.

Previous research has shown that damage to the DNA in sperm may cause infertility or increase the chances of miscarriage, if the damage is extensive (eg. present in the overwhelming majority of sperm). Some studies suggest that DNA damage can be caused by oxidative stress. Antioxidants, such as Vitamin E, which are present in some foods, can prevent damage to cells from "free radicals", which are naturally present by-products of metabolism. We ask whether there is a correlation between sperm DNA damage and Vitamin E

DETAILED DESCRIPTION:
Sperm DNA damage is an emerging cause of male infertility that is likely to be more common among men with increased reactive oxygen species in the ejaculate. Vitamin E can protect the sperm membrane from oxidative damage and increased levels are associated with low levels of reactive oxygen species. This is a study of Vitamin E levels in the spermatozoa and sera of 48 infertile men, and 20 fertile men as a control group, to look for correlations between sperm vitamin E levels and the degree of sperm DNA fragmentation. Dietary intake of antioxidants will also be included.

ELIGIBILITY:
Inclusion Criteria:

* infertile men with previously abnormal semen analyses.
* Control group: fertile adult males

Exclusion Criteria:

* Proxceed use within 3 months of the start of study.
* Vitamin E supplements with > 45 IU daily

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Infertility clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2004-06; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
correlate vitamin E levels in spermatozoa with degree of DNA fragmentation in infertile men

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Lewis, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Department of OB/GYN, Rochester, New York, United States